CLINICAL TRIAL: NCT02227069
Title: A Phase 1, 21-Day, Randomized, Evaluator Blinded, Controlled Study to Evaluate the Irritation Potential of M518101 in Healthy Volunteers, Using a Cumulative Irritant Patch Test Design
Brief Title: Skin Safety Study to Evaluate the Irritation Potential in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maruho North America Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: M518101-US06
Record Dates: First submitted 2014-08-21; First posted 2014-08-27 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Sodium Dodecyl Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- M518101 (Experimental): M518101 is applied topically under occlusive patch conditions to the infrascapular area of the back, once daily for 21 consecutive days over 3 weeks
  Interventions: Drug: M518101
- M518101 Vehicle (Placebo Comparator): M518101 vehicle is applied topically under occlusive patch conditions to the infrascapular area of the back, once daily for 21 consecutive days over 3 weeks
  Interventions: Drug: M518101 Vehicle
- sodium lauryl sulfate (Active Comparator): A solution of 0.2% sodium lauryl sulfate is applied topically under occlusive patch conditions to the infrascapular area of the back once daily for 21 days over 3 weeks, will serve as a positive control.
  Interventions: Other: sodium lauryl sulfate
- Saline (Sham Comparator): A solution of 0.9% saline is applied topically under occlusive patch conditions to the infrascapular area of the back once daily for 21 days over 3 weeks, will serve as a negative control.
  Interventions: Other: saline

INTERVENTIONS:
Drug: M518101
  Arms: M518101
Drug: M518101 Vehicle
  Arms: M518101 Vehicle
Other: sodium lauryl sulfate
  Arms: sodium lauryl sulfate
Other: saline
  Arms: Saline

SUMMARY:
This is a single center, randomized, controlled, within-subject comparison, multiple dose study to determine the irritation potential of M518101 on normal skin under occlusive patch condition.

The study drug will be applied for 21 days under occlusive patch condition. The irritation potential of M518101 will be compared with positive, negative control and M518101 vehicle. The study duration is 21days and there will be at least 23 visits to study center including screening visit.

ELIGIBILITY:
Inclusion Criteria:

* Health male or female subjects age 18 years or older
* Signed and dated Informed Consent Form obtained prior to any study-related activities
* Subjects are free of any systemic or dermatologic disorder
* For Female, females of non-childbearing potential or who agree to use a highly effective method of birth control during the study and have a negative urine pregnancy test.
* Subjects must be able to communicate with the investigator and understand and comply with the requirements of the study and visit schedule

Exclusion Criteria:

* Have any visible skin disease at the application site which will interfere with the evaluation of the test site reaction
* Have damaged skin in or around the test sites
* Have a history of sensitivity to adhesive tape
* Have a known sensitivity to constituents present in the material being evaluated
* Have a history of, or are currently being treated for skin cancer
* have used any study drug and/or participate in any clinical study within 60 days prior to Randomization
* to engage in any type of strenuous exercise (swimming, running, etc.) or who intended to use hot tubs or saunas during the study
* Are pregnant, breastfeeding, or of childbearing potential and who wish to become pregnant during the study
* Are deemed to be ineligible by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Inflammatory skin responses | 21 Days
  Drug application sites will be evaluated for signs of inflammatory skin responses (e.g. erythema, edema, papules) and superficial effects.

CONTACTS AND LOCATIONS:
Locations (1):
- TKL research, Fair Lawn, New Jersey, United States